CLINICAL TRIAL: NCT04295837
Title: A Better Everyday Life - a Complex Intervention Addressing Ability to Perform Activities of Daily Living Among Persons Living With Chronic Conditions
Brief Title: A Better Everyday Life Among Persons With Chronic Conditions
Acronym: ABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Research Institute (Other)
Collaborators: University of Southern Denmark (Other); VIA University College (Other)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, Senior researcher, associate professor, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 145
Record Dates: First submitted 2019-12-05; First posted 2020-03-05 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Chronic Conditions, Multiple
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABLE - A Better everday LifE (Experimental): A home-based occupational therapy intervention addressing ADL task performance issues among persons living with chronic conditions. The ABLE intervention is occupation-focused and -based, and follows a structured process of assessment, goalsetting, intervention and evaluation.
  Interventions: Other: ABLE
- Usual care (Active Comparator): Community-based occupational therapy addressing ADL task performance issues among persons living with chronic conditions
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ABLE — Home-based occupational therapy compensatory programme addressing activities of daily living
  Arms: ABLE - A Better everday LifE
Other: Usual Care — Standard occupational therapy
  Arms: Usual care

SUMMARY:
Background: Persons living with chronic conditions often have decreased ability to perform Activities of Daily Living (ADL) tasks, stressing a need to develop and evaluate intervention programs addressing decreased ADL ability. Guided by the British Medical Research Council's guidance (MRC) on how to develop and evaluate complex interventions, the program "A Better everyday LifE" (ABLE), a home-based intervention program, was developed and feasibility tested. The current phase concerns a full-scale evaluation of the ABLE program including evaluation of effectiveness, processes and cost-effectiveness.

Material and Methods: The design involves a randomized controlled trial, initiated with an internal pilot. The study will include eighty (n=80) home dwelling persons living with chronic conditions, experiencing problems performing ADL. Participants are randomized to either intervention (ABLE) or control (usual care).

Co-primary outcomes are self-reported ADL ability measured using ADL-Questionnaire (ADL-Q) and observed ADL motor ability measured using Assessment of Motor and Process Skills (AMPS). Secondary outcomes are perceived satisfaction with ADL task performance measured using ADL-Q; observed ADL process ability measured using AMPS; and Goal Attainment measured using Goal-Attainment-Scaling (GAS). Data is collected at baseline, post intervention and six months after baseline. Process evaluation data are collected using registration forms and semi-structured qualitative interviews.

The economic evaluation will be performed from a health care sector perspective with 6 months follow-up. Costs will be estimated based on micro costing and national registries. Effects will be Quality Adjusted Life Years and changes in AMPS ADL ability.

DETAILED DESCRIPTION:
Due to the Covid-19 pandemic, the study was truncated on March 11th 2020. Data collected at this time was assessed to be sufficient to answer most pilot study questions, and it was decided to turn the internal pilot into an external pilot. Based on the results of the external pilot, a few adjustments on outcome measurements, inclusion criteria and extraction of information on usual care were applied, before initiation of the full scale trial. Hence ADL-I replaced ADL-Q as primary outcome measurement. Data collection for full scale trial was initiated August 1st 2020.

ELIGIBILITY:
Inclusion Criteria:

* ≥ one year since medical diagnosed with one or more chronic conditions
* Perceive problems performing ADL tasks
* ≥ 18 years of age
* Lives in own home
* Motivated and ready for making changes in ADL performance
* Motivated and ready to participate in program
* Communicates independently and relevant
* Able to understand and relevantly answer a questionnaire

Exclusion Criteria:

* PADL problems with acute need for help (if the client does not already receive help from home carer
* Known substance abuse
* Mental illness, and/or other acute illness effecting ADL task performance
* Communication barriers (e.g. severe cognitive deficits; and barriers that prevents receiving information on study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Change in observed ADL motor ability - with the Assessment of Motor and Process Skills (AMPS) | Week 10
  Observation-based measure of ADL ability - motor
Change in self-reported ADL ability - with the ADL-Interview (ADL-I) | Week 10
  Self-report based on interview addressing perceived ability to perform ADL tasks. Linear measures of ADL ability will be generated using Rasch measurement models. Higher scores mean more ADL ability.

SECONDARY OUTCOMES:
Change in observed ADL process ability - with the Assessment of Motor and Process skills (AMPS) | Week 10
  Observation-based measure of ADL ability - process
Change in observed ADL process ability - with the Assessment of Motor and Process skills (AMPS) | Week 27
  Observation-based measure of ADL ability - process
Change in observed ADL motor ability - with the Assessment of Motor and Process skills (AMPS) | Week 27
  Observation-based measure of ADL ability - motor
Change in self-reported satisfaction with ADL ability - with the ADL-Interview (ADL-IS) | Week 10
  Self-report based on interview addressing satisfaction with perceived ability to perform ADL tasks. Linear measures of satisfactions with ADL ability will be generated using Rasch measurement models. Higher scores mean more satisfaction.
Change in self-reported satisfaction with ADL ability - with the ADL-Interview (ADL-IS) | Week 27
  Self-report based on interview addressing satisfaction with perceived ability to perform ADL tasks. Linear measures of satisfactions with ADL ability will be generated using Rasch measurement models. Higher scores mean more satisfaction.
Change in self-reported ADL ability - with the ADL-Interview (ADL-I) | Week 27
  Self-report based on interview addressing perceived ability to perform ADL tasks. Linear measures of ADL ability will be generated using Rasch measurement models. Higher scores mean more ADL ability.

OTHER OUTCOMES:
Occupational Balance Questionnaire (OBQ11) | Week 10
  Assessing occupational balance
Occupational Balance Questionnaire (OBQ11) | Week 27
  Assessing occupational balance
EuroQoL 5 dimensions (EQ-5D) | Week 10
  Quality of life
EuroQoL 5 dimensions (EQ-5D) | Week 27
  Quality of life
Transition Questionnaire (TRANS-Q) | Week 10
  Perceived change in performance and satisfaction with ADL ability on a Likert scale from much less able/satisfied to fully able/satisfied.
Transition Questionnaire (TRANS-Q) | Week 27
  Perceived change in performance and satisfaction with ADL ability on a Likert scale from much less able/satisfied to fully able/satisfied.
General Health (SF36-SF1) | Week 10
  Perceived general health on 5-point ordinal scale
General Health (SF36-SF1) | Week 27
  Perceived general health on 5-point ordinal scale
Client-Weighted-Problems (CWP) | Week 10
  Self-reported weight of identified problems, need for help and hope for the future on an 11-point ordinal scale ranging from '0' representing "not at all" to '10' representing "to a high extent".
Client-Weighted-Problems (CWP) | Week 27
  Self-reported weight of identified problems, need for help and hope for the future on an 11-point ordinal scale ranging from '0' representing "not at all" to '10' representing "to a high extent".

CONTACTS AND LOCATIONS:
Overall Officials: Eva E Wæhrens, PhD, Principal Investigator — The Parker Research Institute, Bispebjerg and Frederiksberg Hospital
Locations (1):
- The Parker Research Institute, Department of Rheumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hagelskjaer V, Nielsen KT, von Bulow C, Oestergaard LG, Graff M, Waehrens EE. Evaluating a complex intervention addressing ability to perform activities of daily living among persons with chronic conditions: study protocol for a randomised controlled trial (ABLE). BMJ Open. 2021 Nov 26;11(11):e051722. doi: 10.1136/bmjopen-2021-051722. PMID 34836902
- [Derived] Hagelskjaer V, Nielsen KT, von Bulow C, Graff M, Waehrens EE. Occupational therapy addressing the ability to perform activities of daily living among persons living with chronic conditions: a randomised controlled pilot study of ABLE 2.0. Pilot Feasibility Stud. 2021 Jun 11;7(1):122. doi: 10.1186/s40814-021-00861-9. PMID 34116727